

A Social Media Intervention for Exercise Motivation and Cardiac Rehabilitation Adherence 11/08/2018

## **Facebook Study Information Sheet**

A feasibility research study is being done to examine the use of a private Facebook group to deliver information and support for cardiac rehabilitation patients at the Cleveland Clinic.

- The goal of this study is to examine social media and motivation for exercise.
- You are being asked to participate because you are a patient who plans to take part in cardiac rehabilitation at Cleveland Clinic and you are a current Facebook user.

There are no known risks associated with this study, however, due to the social nature of Facebook, comments made will be seen by the study staff and by other participants in the private group.

Confidentiality is always a concern with research. To protect the confidentiality and privacy of the patients who participate in the Facebook study, your information and participation in this study will be kept confidential. All data will be stored in a locked file cabinet in the investigator's locked office.

### What is involved if you decide to take part in this study?

As part of this study you will be assigned to either a Facebook group or a comparison group. This will be done randomly, like a flip of the coin. Neither the principal investigator nor the participant can choose to which group they will be assigned.

At the start of the study, you will be asked to fill out 2 questionnaires called the BREQ-3 and PNSE. These will take about 10 minutes and will appear at the end of this information sheet. If you are assigned to the Facebook group, you will be given information for joining private Facebook group for cardiac rehabilitation. You will receive information and be able to talk with other cardiac rehabilitation patients on the Facebook group.

If you are randomized to the comparison group you will receive the same educational information via email.

The information that you receive will be in addition to what you receive at your cardiac rehabilitation sessions. You will receive the same care in cardiac rehabilitation regardless of which group you are randomized.

When you are done with cardiac rehabilitation you will be asked to fill out the BREQ-3 and the PNSE again as well as an anonymous questionnaire about your experience with the Facebook group.

Information for this study will be collected from Facebook, from the medical record, and from the BREQ-3 and the PNSE.

Results of this study will be shared through publication and presentations. No personal or identifiable information will be shared.

#### **Future Research:**

Facebook Information Sheet V1 11/8/18

Content from postings/conversations on the Facebook group may be used for future research.

Comments from the questionnaire will help the researchers determine if a larger study is feasible.

Your participation in this study will last 12 weeks. Thereafter, you may continue to access the Facebook group. If you have been randomized to the comparison group, you will be able to access the Facebook group at the end of 12 weeks.

# What are possible benefits of participating in the research?

You may or may not benefit directly from participation in this study. The knowledge gained from this study may benefit future patients.

## Are there any costs to you if you participate in this study?

There will be no cost to any participant as part of this study.

The services that you receive as part of conventional routine care in cardiac rehabilitation will be billed to you or your health insurance plan. You are responsible for paying any deductibles, copayments or co-insurance that are a normal part of your health insurance plan.

## Are there any payments to you if you participate in this study?

You will receive no payment or compensation if you volunteer for this study.

## What will happen to your information that is collected for this research?

Cleveland Clinic has rules and procedures to protect information about you. Federal and State laws also protect your privacy.

The research team working on the study will collect information about you. This includes your health information, data collected for this research study and personal identifying information including your name, address, date of birth and other identifying information.

Generally, only people on the research team will know your identity and that you are in the research study. However, sometimes other people at Cleveland Clinic may see or give out your information. These include people who review research studies including the Institutional Review Board and Research Compliance, their staff, lawyers, or other Cleveland Clinic staff.

People outside Cleveland Clinic may need to see your information for this study. Examples include government groups (such as the Food and Drug Administration), safety monitors, other hospitals in the study and the sponsor of the research and their agents. Cleveland Clinic will do our best to ensure your information is kept confidential and that only the health information which is minimally required to conduct the study is used or disclosed to people outside Cleveland Clinic; however, people outside Cleveland Clinic who receive your information may not be covered by this promise.

You do not have to give this permission to use and give out your information; however you will not be able to participate in this research study without providing this permission by signing this consent form. The use and disclosure of your information has no expiration date.

Facebook Information Sheet V1 11/8/18

You may cancel your permission to use and disclose your information at any time by notifying the Principal Investigator in writing:

Lee Anne Siegmund PhD, RN 9500 Euclid Ave. P3-206A Cleveland, Ohio 44195.

If you do cancel your permission to use and disclose your information, your participation in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in the study.

Your decision to participate is completely voluntary and will have no effect on the quality of your medical care if you choose not to participate. You can also withdraw from the study at any time. Your decision to participate or not, will not impact your nursing or medical care.

If you have any questions or concerns about this study contact Lee Anne Siegmund PhD, RN at (216) 445-3457. If you have questions about your rights as a research participant, contact the Institutional Review Board at (216) 444-2914.

Completion of the questionnaires that follow indicates your agreement to participate in the study.